CLINICAL TRIAL: NCT05132127
Title: An Open-label Study for Sutimlimab in Participants With Cold Agglutinin Disease (CAD) Who Have Completed the CARDINAL Study (BIVV009-03/EFC16215, Part B) or CADENZA Study (BIVV009-04/EFC16216, Part B) in Japan
Brief Title: Sutimlimab (BIVV009) for the Adult Participants With Cold Agglutinin Disease (CAD) Who Have Completed Phase 3 Studies (CARDINAL or CADENZA) in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17352; U1111-1266-5421 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cold Agglutinin Disease
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — sutimlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sutimlimab (Experimental): Participants with body weight greater than or equal to (>=) 39 kilograms (kg) to less than (<) 75 kg and who had completed Part B of CARDINAL or CADENZA study were enrolled in the current study and received sutimlimab (BIVV009) 6.5 grams as intravenous (IV) infusion on Day 0, Day 7, Day 21 and thereafter every 2 weeks (maximum duration: 49 weeks) in the current study.
  Interventions: Drug: sutimlimab

INTERVENTIONS:
Drug: sutimlimab — Pharmaceutical form: solution for injection Route of administration: intravenous (IV)

SUMMARY:
This was a multi-center, single treatment-group, open-label study to provide sutimlimab to the adult participants with cold agglutinin disease (CAD) who had completed the CARDINAL (NCT number: NCT03347396) or CADENZA (NCT number: NCT03347422) studies and benefitted from sutimlimab treatment in Japan.

• Study and treatment duration: the period between the participant's completion of the CARDINAL and CADENZA studies and sutimlimab or other appropriate CAD therapy becoming commercially available to participants in Japan.

DETAILED DESCRIPTION:
The period between screening/baseline visit (upon the participant's completion* of the CARDINAL and CADENZA studies) and end of treatment with sutimlimab in this study was determined by sutimlimab or other appropriate CAD therapy becoming commercially available to participants in Japan.

ELIGIBILITY:
Inclusion Criteria:

--Participant must be adults.

* Participants who had been enrolled in and had completed Part B of CARDINAL or CADENZA study.
* Participants who had ongoing diagnosis of CAD.
* Participants who continued to require treatment for CAD upon completion of participation in the previous study evidenced by return of CAD-related symptoms of anemia and/or deterioration on markers of hemolysis after the end of study visit following the 9-week safety follow up period. (9-week follow up period).
* Participants who had acceptable benefit/risk profile.
* Participant who had acceptable infection risk.
* Participants who had no available appropriate alternative therapy for CAD.
* Body weight >= 39 kg.
* Gave signed informed consent.

Exclusion Criteria:

--Clinical diagnosis of systemic lupus erythematosus or immune complex-mediated autoimmune disorders.

* Participants who met recent Rituximab and/or immunosuppressive therapy.
* Any of the following medical conditions:

  1. Active, serious intercurrent illness which precluded enrolment until recovery was complete.
  2. Pregnancy or breast-feeding.
* End of Study visit in CARDINAL or CADENZA took place more than 3 months before Baseline visit in this study.
* Hypersensitivity reactions to sutimlimab or components thereof, or other allergy that, in the opinion of the Investigator, contraindicated participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Japan (5):
  - Investigational Site Number 3920005, Ishikawa
  - Investigational Site Number 3920004, Kanagawa
  - Investigational Site Number 3920003, Osaka
  - Investigational Site Number 3920002, Saitama
  - Investigational Site Number 3920001, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17352 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25303&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 active sites in Japan. A total of 7 participants were enrolled from 11 November 2021 to 07 December 2021. Participants with cold agglutinin disease (CAD) and who had completed Part B of CARDINAL (NCT03347396) or CADENZA (NCT03347422) study and benefitted from sutimlimab treatment were enrolled in the current study.
Pre-assignment Details: Per protocol, enrolled participants were planned to receive sutimlimab based on their baseline body weight as: 6.5 grams for baseline body weight of greater than or equal to (>=) 39 kilograms (kg) to less than (<) 75 kg or 7.5 grams for baseline body weight of >= 75 kg. As no participant had a Baseline body weight >= 75 kg, per the study protocol, 7.5 grams dose was not administered.
Groups:
- Sutimlimab: Participants with body weight >= 39 kg to < 75 kg and who had completed Part B of CARDINAL or CADENZA study were enrolled in the current study and received sutimlimab (BIVV009) 6.5 grams as intravenous (IV) infusion on Day 0, Day 7, Day 21 and thereafter every 2 weeks (maximum duration: 49 weeks) in the current study.
Period: Overall Study
Arm/Group | Sutimlimab
Started | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all enrolled participants who took at least 1 dose of study intervention.
Groups:
- Sutimlimab: Participants with body weight >= 39 kg to < 75 kg and who had completed Part B of CARDINAL or CADENZA study were enrolled in the current study and received sutimlimab (BIVV009) 6.5 grams as IV infusion on Day 0, Day 7, Day 21 and thereafter every 2 weeks (maximum duration: 49 weeks) in the current study.
Arm/Group | Sutimlimab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study intervention and did not necessarily had to have a causal relationship with the treatment. Serious adverse events (SAEs) were defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/ incapacity, was a congenital anomaly/birth defect, suspected transmission of any infectious agent via an authorized medicinal product, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent period (from first dose of study intervention up to 9 weeks after the last dose of study intervention in the current study).
Time Frame: From first dose of study intervention up to 9 weeks after the last dose of study intervention (maximum duration: 49 weeks)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sutimlimab
Number analyzed (Participants) | 7
Participants
  TEAEs | 7
  TESAEs | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (AESI)
Description: An AE was defined as any untoward medical occurrence in a participant who received study intervention and did not necessarily had to have a causal relationship with the treatment. AESIs were AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the investigator to the Sponsor was required.
Time Frame: as for outcome 1
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sutimlimab
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of study intervention up to 9 weeks after the last dose of study intervention (maximum duration: 49 weeks)
Description: Analysis was performed on safety population.
Arm/Group | Sutimlimab
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sutimlimab (N=7)
Spontaneous Bacterial Peritonitis (Infections and infestations) | 1 (1)
Cholangitis Acute (Hepatobiliary disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sutimlimab (N=7)
Cystitis (Infections and infestations) | 1 (2)
Gingivitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Skin Candida (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (9)
Lip Haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Epidermolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Vaccination Site Pain (General disorders) | 1 (2)
Blood Immunoglobulin M Increased (Investigations) | 1 (1)
Blood Iron Decreased (Investigations) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1)
Cytomegalovirus Test Positive (Investigations) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT05132127/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05132127/SAP_001.pdf